CLINICAL TRIAL: NCT06063967
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy and Safety of Risankizumab Subcutaneous Induction Treatment in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Risankizumab Subcutaneous Induction Treatment for Moderately to Severely Active Crohn's Disease.
Acronym: AFFIRM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M23-784; 2024-516023-13-00 (Other: EU CT)
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease
Keywords: Risankizumab, Skyrizi, Crohn's Disease, ABBV-066
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Period A: Risankizumab Dose A (Experimental): Participants randomized to receive risankizumab Dose A administered by subcutaneous (SC) injection for up to 12 weeks during Period A.
  Interventions: Drug: Risankizumab SC
- Period A: Placebo (Placebo Comparator): Participants randomized to receive placebo for risankizumab administered by Subcutaneous (SC) injection for up to 12 weeks during Period A.
  Interventions: Drug: Placebo for risankizumab
- Period B: Risankizumab Dose B (Experimental): Participants randomized to receive risankizumab Dose A in Period A that achieved adequate response to receive risankizumab Dose B administered by subcutaneous (SC) injection for up to 12 weeks.
  Interventions: Drug: Risankizumab SC
- Period B: Placebo (Placebo Comparator): Participants randomized to receive placebo risankizumab in Period A that achieved adequate response to continue to receive placebo for risankizumab administered by Subcutaneous (SC) injection for up to 12 weeks in Period B.
  Interventions: Drug: Placebo for risankizumab
- Period B: Risankizumab Dose C (Experimental): Participants with inadequate response in Period A to receive Dose C administered by Subcutaneous (SC) injection for up to 12 weeks during Period B.
  Interventions: Drug: Risankizumab SC
- Period C: Open-Label Risankizumab Dose D (Experimental): Participants who complete the Period B Week 24 visit to receive open-label risankizumab Dose D administered by subcutaneous (SC) injection for up to 52 weeks during Period C.
  Interventions: Drug: Risankizumab SC

INTERVENTIONS:
Drug: Risankizumab SC — subcutaneous (SC) injection
  Other Names: ABBV-066; SKYRIZI
  Arms: Period A: Risankizumab Dose A; Period B: Risankizumab Dose B; Period B: Risankizumab Dose C; Period C: Open-Label Risankizumab Dose D
Drug: Placebo for risankizumab — subcutaneous (SC) injection
  Arms: Period A: Placebo; Period B: Placebo

SUMMARY:
Crohn's disease (CD) is a long-lasting disease that causes severe inflammation (redness, swelling), in the digestive tract, most often affecting the bowels. It can cause many different symptoms including abdominal pain, diarrhea, tiredness, and weight loss. This study will assess how safe and effective risankizumab subcutaneous (SC) induction treatment is in treating moderately to severely active CD in adult participants.

Risankizumab is an approved drug for adults with CD. This study comprises of a Period A, a Period B, and a Period C. In Period A, participants are placed in 1 of 2 groups to receive either risankizumab SC Dose A or Placebo. In Period B, based on response, participants will receive risankizumab SC Dose B or Placebo. Participants who do not have improvement in CD symptoms at Week 12 will receive risankizumab SC Dose C and participants with worsening CD symptoms in period B will receive risankizumab SC. In Period C, eligible participants will receive open-label risankizumab SC Dose D. Approximately 276 adult participants with a diagnosis of moderately to severely active CD will be enrolled in approximately 250 sites globally.

Participants will receive SC induction treatment of risankizumab or matching placebo for up to 24 weeks in Period A and B followed by an open-label risankizumab extension in Period C for 52 weeks. The duration of the study will be approximately 93 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed diagnosis of CD for at least 3 months prior to Baseline.
* Participant meets the following disease activity criteria:

  1. Moderate to severe CD as assessed by CDAI
  2. Endoscopic evidence of mucosal inflammation as documented by a SES-CD
* Participant has demonstrated intolerance, loss of response or inadequate response to conventional or advanced therapies for CD.

Exclusion Criteria:

* Participants with a current diagnosis of ulcerative colitis or indeterminate colitis.
* Participants with unstable doses of concomitant Crohn's disease therapy.
* Participants with prior exposure to p19 inhibitors.
* Participants with complications of Crohn's disease.
* Participants having an ostomy or ileoanal pouch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Remission (CDAI < 150) | Week 12
  The CDAI consists of 8 components; 7 are based on participant diary entries, participant interviews, physical examinations, measurement of body weight and height and 1 is based on laboratory analysis. CDAI clinical remission of Crohn's disease is defined as CDAI < 150
Percentage of Participants With Endoscopic Response | Week 12
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline)
Number of Participants Experiencing Adverse Events | Up to approximately 96 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Remission | Week 12
  Clinical remission is defined as using the average daily Stool Frequency (SF) ≤ 2.8 and not worse than Baseline AND average daily Abdominal Pain (AP) score ≤ 1 and not worse than Baseline.
Percentage of Participants With Endoscopic Remission | Week 12
  Endoscopic remission: SES-CD ≤ 4 and at least a 2 point reduction versus baseline and no subscore greater than 1 in any individual variable
Percentage of Participants With Ulcer-Free Endoscopy | Week 12
  Ulcer-free endoscopy: SES-CD ulcerated surface subscore of 0 in participants with SES-CD ulcerated surface subscore ≥ 1 at Baseline
Change From Baseline of Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue | Week 12
  The FACIT-Fatigue scale is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a 5-point Likert scale. The FACIT Fatigue Scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better the quality of life. A positive change from baseline indicates improvement.
Percentage of Participants with a CR-100 Clinical Response | Week 4
  CR-100 defined as at least a 100-point reduction from Baseline in CDAI

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (179):
- United States (79):
  - Gi Alliance - Arizona Digestive Health - Sun City /ID# 268178, Sun City, Arizona
  - Kindred Medical Institute - Corona /ID# 262075, Corona, California
  - Southern California Res. Ctr. /ID# 256612, Coronado, California
  - Valley Clinical Trials, LLC dba Flourish Research /ID# 256610, Covina, California
  - Newport Huntington Medical Group /ID# 256622, Huntington Beach, California
  - Om Research LLC /ID# 259645, Lancaster, California
  - Om Research LLC /ID# 267523, Lancaster, California
  - Clinnova Research - Orange /ID# 270138, Orange, California
  - University of California, Irvine Medical Center /ID# 259677, Orange, California
  - Prospective Research Innovations Inc. /ID# 267856, Rancho Cucamonga, California
  - University of California San Francisco - Mission Bay /ID# 267529, San Francisco, California
  - Amicis Research Center - Valencia /ID# 269158, Valencia, California
  - OM Research LLC /ID# 268735, Victorville, California
  - Danbury Hospital, Western Connecticut Health Network /ID# 261851, Danbury, Connecticut
  - Novum Research /ID# 269223, Clermont, Florida
  - Research Associates of South Florida, LLC /ID# 261627, Coral Gables, Florida
  - University of Florida College of Medicine /ID# 261248, Gainesville, Florida
  - Auzmer Research /ID# 261437, Lakeland, Florida
  - Cfagi Llc /Id# 262005, Maitland, Florida
  - Atlantic Medical Research /ID# 256471, Margate, Florida
  - Homestead Associates in Research /ID# 259643, Miami, Florida
  - University of Miami /ID# 256587, Miami, Florida
  - JD Medical Group, LLC /ID# 262185, Miami, Florida
  - Gastroenterology Group Naples /ID# 256566, Naples, Florida
  - Sarkis Clinical Trials - Ocala /ID# 267840, Ocala, Florida
  - Endoscopic Research, Inc. /ID# 256597, Orlando, Florida
  - AdventHealth Medical Group Blood & Marrow Transplant at Orlando /ID# 261811, Orlando, Florida
  - GCP Clinical Research, LLC /ID# 260342, Tampa, Florida
  - Avita Clinical Research /ID# 261640, Tampa, Florida
  - Winship Cancer Institute of Emory University /ID# 261877, Atlanta, Georgia
  - Mount Vernon Clinical Research /ID# 271813, Atlanta, Georgia
  - Atlanta Ctr. for Gastro /ID# 261181, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 256611, Macon, Georgia
  - Gastroenterology Consultants, P.C /ID# 260635, Roswell, Georgia
  - Grand Teton Research Group /ID# 267521, Idaho Falls, Idaho
  - Duplicate_The University of Chicago DCAM /ID# 256577, Chicago, Illinois
  - GI Alliance - Glenview /ID# 257744, Glenview, Illinois
  - GI Alliance - Gurnee /ID# 257735, Gurnee, Illinois
  - Southwest Gastroenterology /ID# 256619, Oak Lawn, Illinois
  - IU Health University Hospital /ID# 259633, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 262551, Kansas City, Kansas
  - Cotton O'Neil Clinical Research Center, Digestive Health /ID# 256592, Topeka, Kansas
  - University of Louisville Hospital /ID# 256569, Louisville, Kentucky
  - Louisiana Research Center, LLC /ID# 256598, Shreveport, Louisiana
  - Portland Gastroenterology Center - Portland - Congress Street /ID# 268428, Portland, Maine
  - Massachusetts General Hospital /Id# 261051, Boston, Massachusetts
  - Clin Res Inst of Michigan, LLC /ID# 256609, Chesterfield, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 261017, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 256568, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 256594, Rochester, Minnesota
  - Saint Lukes Hospital of Kansas City /ID# 271816, Kansas City, Missouri
  - Allied Health Clinical Research Organization, LLC /ID# 261618, Englewood, New Jersey
  - NY Scientific /ID# 261209, Brooklyn, New York
  - Columbia University Medical Center /ID# 261879, New York, New York
  - New York Gastroenterology Associates /ID# 257730, New York, New York
  - Univ NC Chapel Hill /ID# 256368, Chapel Hill, North Carolina
  - Carolina Research /ID# 261435, Greenville, North Carolina
  - Boice-Willis Clinic, P.A. /ID# 262209, Rocky Mount, North Carolina
  - Plains Clinical Research Center, LLC /ID# 256602, Fargo, North Dakota
  - Optimed Research, Ltd. /ID# 256573, Columbus, Ohio
  - The Ohio State University - Hilliard /ID# 256623, Hilliard, Ohio
  - Hightower Clinical /ID# 256613, Oklahoma City, Oklahoma
  - Options Health Research /ID# 271243, Tulsa, Oklahoma
  - Gastro One /ID# 256614, Cordova, Tennessee
  - Quality Medical Research /ID# 262077, Nashville, Tennessee
  - Amel Med LLC. /ID# 259642, Austin, Texas
  - Novel Research - Bellaire /ID# 269788, Bellaire, Texas
  - University of Texas - Southwestern Medical Center /ID# 268157, Dallas, Texas
  - Digestive Health Associates of Texas (DHAT) Research Institute - Garland /ID# 256596, Garland, Texas
  - Baylor College of Medicine /ID# 256600, Houston, Texas
  - LinQ Research /ID# 267880, Houston, Texas
  - GI Alliance/TDDC /ID# 261623, Lubbock, Texas
  - North Hills Medical Research - North Richard Hills /ID# 268411, North Richland Hills, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 256599, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 256601, San Antonio, Texas
  - Tyler Research Institute, LLC /ID# 256595, Tyler, Texas
  - GI Alliance Bay Area Gastroenterology /ID# 261866, Webster, Texas
  - University Physicians and Surgeons Inc. /ID# 259636, Huntington, West Virginia
  - Wisconsin Center for Advanced Research /ID# 256575, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Britanico de Buenos Aires /ID# 256011, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Gedyt /ID# 258984, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 256690, Córdoba
- Brazil (6):
  - L2ip - Instituto De Pesquisas Clínicas /ID# 261491, Brasília, Federal District
  - Galileo Medical Research Ltda /ID# 261493, Juiz de Fora, Minas Gerais
  - Hospital de Clinicas de Porto Alegre /ID# 261496, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 261490, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 261489, Ribeirão Preto, São Paulo
  - Rocco & Nazato Servicos Medicos /ID# 261497, São Paulo, São Paulo
- Canada (5):
  - University of Calgary /ID# 264640, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 261155, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre - Victoria General /ID# 257072, Halifax, Nova Scotia
  - Toronto Digestive Disease Associates /ID# 260532, Vaughan, Ontario
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 262179, Montreal, Quebec
- Chile (7):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 256398, Concepción, Bio-Bio
  - Sociedad de Servicios Medicos Walsen Galmez Ltda. /ID# 256397, Providencia, Region Metropolitana Santiago
  - Centros Medicos Espacioeme Spa /Id# 262844, Santiago, Region Metropolitana Santiago
  - Pontificia Universidad Catolica de Chile /ID# 256935, Santiago, Region Metropolitana Santiago
  - Serv Salud Metropolitano Central Hospital Clinico San Borja Arriaran /Id# 260765, Santiago, Region Metropolitana Santiago
  - Clinica Dermacross /ID# 260769, Vitacura, Region Metropolitana Santiago
  - Hospital Clinico Universidad De Los Andes /ID# 256856, Santiago
- China (16):
  - Chongqing General Hospital /ID# 260941, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University /ID# 260944, Xiamen, Fujian
  - Guangzhou First People's Hospital /ID# 260943, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 260248, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 260247, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University /ID# 261281, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University /ID# 260938, Changsha, Hunan
  - Changzhou No.2 Peoples Hospital /ID# 260935, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital /ID# 260942, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 260934, Nanjing, Jiangsu
  - Wuxi PeopleS Hospital /ID# 270166, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 260936, Nanchang, Jiangxi
  - Renji Hospital, Shanghai Jiaotong University School Of Medicine /ID# 270165, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 260251, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine /ID# 260246, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Henan University of Science and Technology /ID# 260933, Luoyang
- Czechia (2):
  - Fakultni Thomayerova nemocnice /ID# 272944, Prague, Praha 4
  - Nemocnice Ceske Budejovice a.s. /ID# 256414, České Budějovice
- Hungary (3):
  - Duplicate_Clinfan Szolgaltato Kft. /ID# 260032, Szekszárd, Tolna County
  - Semmelweis Egyetem /ID# 260030, Budapest
  - Semmelweis Egyetem /ID# 274289, Budapest
- Israel (3):
  - Shaare Zedek Medical Center /ID# 256253, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 256251, Ramat Gan, Tel Aviv
  - Bnai Zion Medical Center /ID# 264457, Haifa
- Japan (5):
  - Gamagori City Hospital /ID# 261372, Gamagori-shi, Aichi-ken
  - Tsujinaka Hospital - Kashiwanoha /ID# 261370, Kashiwa-shi, Chiba
  - Hyogo Medical University Hospital /ID# 261371, Nishinomiya-shi, Hyōgo
  - Hamamatsu University Hospital /ID# 268612, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 261373, Sunto-gun, Shizuoka
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 269630, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 269628, Vilnius
- Poland (3):
  - CenterMed Krakow Sp. z o.o. /ID# 273038, Krakow, Lesser Poland Voivodeship
  - Panstwowy Instytut Medyczny MSWiA /ID# 273024, Warsaw, Masovian Voivodeship
  - WSD MEDI Clinical Sp. z o.o. /ID# 273053, Warsaw, Masovian Voivodeship
- Puerto Rico (2):
  - Caribbean Medical Research Center /ID# 268398, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 262250, San Juan
- Saudi Arabia (4):
  - King Fahad Specialist Hospital /ID# 264441, Dammam
  - King Abdulaziz Medical City- National Guard Hospital /ID# 264542, Riyadh
  - King Saud University /ID# 264536, Riyadh
  - King Faisal Specialist Hospital and Research Center /ID# 264539, Riyadh
- Serbia (7):
  - Clinical Hosp Center Zvezdara /ID# 256727, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 256904, Belgrade, Beograd
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 256844, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 257899, Belgrade, Beograd
  - General Hospital Leskovac /ID# 261812, Leskovac, Jablanicki Okrug
  - Opsta Bolnica Pancevo /ID# 266881, Pančevo, Vojvodina
  - University Clinical Center Vojvodina /ID# 256843, Novi Sad
- South Korea (9):
  - Inje University Haeundae Paik Hospital /ID# 268081, Busan, Busan Gwang Yeogsi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 259257, Daejeon, Daejeon Gwang Yeogsi
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 268080, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 262248, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 259255, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 270780, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 259254, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Chilgok Hospital /ID# 262449, Daegu
  - Yonsei University Health System Severance Hospital /ID# 259256, Seoul
- Taiwan (6):
  - National Taiwan University Hospital /ID# 256891, Taipei City, Taipei
  - Show Chwan Memorial Hospital /ID# 272483, Changhua
  - Chiayi Chang Gung Memorial Hospital /ID# 272484, Chiayi City
  - Far Eastern Memorial Hospital /ID# 256893, New Taipei City
  - China Medical University Hospital /ID# 256890, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 256892, Taoyuan
- Turkey (Türkiye) (7):
  - Gazi Universitesi Tip Fakultes /ID# 259747, Yenimahalle, Ankara
  - Kocaeli University Research and Application Hospital /ID# 259750, Dilovası, Kocaeli
  - Ankara City Hospital /ID# 261906, Ankara
  - Antalya Egitim Ve Arastirma Hastanesi /ID# 259746, Antalya
  - Ege University Medical Faculty /ID# 259749, Izmir
  - Dokuz Eylul University Medical Faculty /ID# 262041, Izmir
  - Mersin University Medical /ID# 259748, Mersin
- United Arab Emirates (2):
  - Burjeel Medical City /ID# 269671, Abu Dhabi
  - Sheikh Shakhbout Medical City /ID# 269680, Abu Dhabi
- United Kingdom (8):
  - Velocity Clinical Research Ltd /ID# 271687, High Wycombe, Buckinghamshire
  - Addenbrookes Hospital /ID# 256735, Cambridge, Cambridgeshire
  - St George University Hospitals NHS Foundation Trust /ID# 256729, London, Greater London
  - Velocity North London /ID# 271900, North Finchley, Greater London
  - University Hospitals Birmingham NHS Foundation Trust /ID# 256738, Birmingham
  - The Dudley Group NHS Foundation Trust /ID# 258681, Dudley
  - Whiston Hospital /ID# 261449, Prescot
  - Stepping Hill Hospital /ID# 259867, Stockport

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-784